CLINICAL TRIAL: NCT06273020
Title: The Effect of Cerebrolysin on the Blood-brain-barrier in Patients With Diabetes and Ischemic Stroke
Brief Title: Effect of Cerebrolysin on the Blood Brain Barrier in Patients With Diabetes and Ischemic Stroke
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Ever Neuro Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Juan Fernando Góngora Rivera, MD, PhD, Dr.med. Juan Fernando Góngora Rivera, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MI22-00013
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke, Acute; Diabetes Mellitus, Type 2; Blood Brain Barrier
Keywords: stroke; diabetes mellitus type 2
MeSH Terms: conditions — Ischemic Stroke; Diabetes Mellitus, Type 2; Stroke | interventions — cerebrolysin

STUDY DESIGN:
Intervention Model Description: There are 3 groups in this clinical trial
  Group 1: 20 patients with previous intravenous thrombolysis (IVT) in the qualifying stroke and who agreed to receive and got selected (through randomization) cerebrolysin.
  Group 2 : 20 patients with previous IVT in the qualifying stroke and who agreed to receive cerebrolysin but they were not choose through randomization.
  Group 3: 20 patients that they were not candidates to receive IVT (out of therapeutic window) but agreed to receive cerebrolysin (randomization not used)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous thrombolysis and cerebrolysin (Experimental): Group 1: 20 patients with previous intravenous thrombolysis (IVT) in the qualifying stroke and who agreed to receive and got selected (through randomization) cerebrolysin.
  Cerebrolysin would be prepared according to manufacturer's instructions: 30 mL of cerebrolysin in 100 ml of saline solution every 24 hours to a minimum of 10 days and a maximum of 14 days
  Interventions: Drug: Cerebrolysin; Procedure: Brain-MRI with contrast after 10-14 days of cerebrolysin
- Intravenous thrombolysis without cerebrolysin (Active Comparator): Group 2 : 20 patients with previous IVT in the qualifying stroke and who agreed to receive cerebrolysin but they were not choose through randomization.
  Interventions: Procedure: Brain-MRI with contrast after 10-14 days of cerebrolysin
- Patients with cerebrolysin without IVT (Other): Group 3: 20 patients that they were not candidates to receive IVT (out of therapeutic window) but agreed to receive cerebrolysin (randomization not used)
  Cerebrolysin would be prepared according to manufacturer's instructions: 30 mL of cerebrolysin in 100 ml of saline solution every 24 hours to a minimum of 10 days and a maximum of 14 days
  Interventions: Drug: Cerebrolysin; Procedure: Brain-MRI with contrast after 10-14 days of cerebrolysin

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin would be prepared according to manufacturer's instructions: 30 mL of cerebrolysin in 100 ml of saline solution every 24 hours to a minimum of 10 days and a maximum of 14 days
  Arms: Intravenous thrombolysis and cerebrolysin; Patients with cerebrolysin without IVT
Procedure: Brain-MRI with contrast after 10-14 days of cerebrolysin — Blood-brain barrier (BBB) disruption will be measured using dynamic susceptibility contrast (DSC) magnetic resonance imaging. DSC MRI is collected during the injection of a gadolinium bolus and the majority of the change in recorded signal in this T2-weighted sequence is due to intravascular contrast. However, in the setting of gadolinium leakage through the BBB into the brain parenchyma, the recorded signal is altered by a T1 effect. An arrival time correction is performed to account for regional difference in blood flow after which the signal is separated into an intravascular and an extravascular component using a comparison with unaffected tissue.The extravascular component is captured with the metric K2 which reflects the fraction of the recorded signal that is due to gadolinium leakage and is a measure of BBB disruption.

SUMMARY:
A prospective, single-center study would be carried out in the Neurology Department of the University Hospital "Dr. José Eleuterio González" in order to analyze the effect of cerebrolysin on the blood-brain-barrier in patients with ischemic stroke with personal history of type-2 diabetes

DETAILED DESCRIPTION:
A prospective, single-center study would be carried out in the Neurology Department of the University Hospital "Dr. José Eleuterio González" in order to analyze the effect of cerebrolysin on the blood-brain-barrier (BBB) in patients with ischemic stroke (IS) of the middle cerebral artery with personal history of type-2 diabetes (T2D).

The main objective is to compare the effect of cerebrolysin on the BBB in the above mentioned patients with intravenous thrombolysis (IVT) and without IVT.

The hypothesis of this study is that cerebrolysin can affect the BBB permeability after 10 days of the administration of this drug

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 years.
2. Clinical and imaging criteria for ischemic stroke of the middle cerebral artery.
3. Acute non-lacunar cerebral infarction.
4. Cerebral infarction with a score on the NIH scale between 5 and 20 points.
5. Patient with a previous diagnosis of type 2 diabetes mellitus, regardless of the form of diagnosis, time of evolution, previous or current treatment, adherence or not to treatment, presence or absence of microvascular and/or macrovascular complications.
6. mRs ≤ 1 before the qualifying stroke (functionally independent for all activities of daily living).
7. The patient and/or legal representative or direct family member has signed the informed consent form.

Exclusion Criteria:

1. Advanced disease or terminal with life expectancy < 6 months.
2. - Over 80 years old
3. Lacunar infarction or small vessel disease.
4. Pre-existing medical, neurological, or psychiatric disease that would confound neurological or functional evaluations (eg, Alzheimer's disease, vascular dementia, Parkinson's disease, demyelinating disease, encephalopathy of any cause, history of significant alcohol or drug abuse).
5. Pregnancy or lactation.
6. Acute or chronic renal failure with creatinine clearance <30 mL/min.
7. Allergy or any condition that represents a contraindication for the administration of Cerebrolysin.
8. Treatment with another investigational drug within the past 30 days that may interfere with the study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood-Brain-Barrier Permeability after 10-14days of cerebrolysin in patients with AIS of the middle cerebral artery | After 10-14 days of cerebrolysin
  Blood-brain barrier (BBB) disruption will be measured using dynamic susceptibility contrast (DSC) magnetic resonance imaging (MRI).DSC MRI is collected during the injection of a gadolinium bolus and the majority of the change in recorded signal in this T2*-weighted sequence is due to intravascular contrast. However, in the setting of gadolinium leakage through the BBB into the brain parenchyma, the recorded signal is altered by a T1 effect. An arrival time correction is performed to account for regional difference in blood flow after which the signal is separated into an intravascular and an extravascular component using a comparison with unaffected tissue. The extravascular component is captured with the metric K2 which reflects the fraction of the recorded signal that is due to gadolinium leakage and is a measure of BBB disruption.

SECONDARY OUTCOMES:
Comparison of clinical severity, using NIH Stroke Scale in patients with and withouth cerebrolysin | After 10-14 days of cerebrolysin, and 30 days and 90days after hospital discharge
  The NIH Stroke Scale would be measured in all patients in the indicated time frames, and the results would be compared based among the 3 groups
Comparison of functional prognosis, using modified Rankin scale in patients with and withouth cerebrolysin | After 10-14 days of cerebrolysin, and 30 days and 90days after hospital discharge
  The modified Rankin scale would be measured in all patients in the indicated time frames, and the results would be compared based among the 3 groups
Comparison of cognitive impairment, using Montreal Cognitive Assessment in patients with and withouth cerebrolysin | fter 10-14 days of cerebrolysin, and 30 days and 90days after hospital discharge
  The Montreal Cognitive Assessment would be measured in all patients in the indicated time frames, and the results would be compared based among the 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Góngora-Rivera, Ph.D., Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Servicio de Neurología del Hospital Universitario "Dr.José E. González", Nuevo León, Monterrey, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data would be shared upon reasonable request after the publication of this trial in an indexed journal
Supporting Information: Study Protocol
Time Frame: Anytime after the publication of this trial in an indexed journal
Access Criteria: Design of meta-analysis When in doubt of the veracity of the data